CLINICAL TRIAL: NCT00131274
Title: A Double-Blind, Placebo-Controlled, Randomized Study of the Efficacy (Gleevec Imatinib Mesylate) in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Gleevec Idiopathic Pulmonary Fibrosis (IPF) Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daniels, Craig E., M.D. (Individual)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: CST1571E2401
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2005-10-05 (Estimated); Status verified 2005-08

CONDITIONS: Idiopathic Pulmonary Fibrosis; Lung Disease; Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Respiratory Diseases; Interstitial Lung Disease; Usual Interstitial Pneumonia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases; Pulmonary Fibrosis; Respiratory Tract Diseases; Lung Diseases, Interstitial | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate (Gleevec)

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Gleevec (imatinib mesylate) in the treatment of idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
This is a multicenter, double-blind, parallel, placebo-controlled, randomized phase 2 study to evaluate the safety and efficacy of Gleevec (imatinib mesylate) in the treatment of Idiopathic Pulmonary Fibrosis (IPF). One-hundred- twenty patients will be enrolled in the trial in total. Subjects must have a diagnosis made by HRCT showing definite or probable IPF and clinical symptoms consistent with IPF with onset between 3 and 36 months prior to screening. Subjects will be randomly assigned to receive either Gleevec 600 mg orally or placebo, once per day for approximately 2 years. The primary efficacy will be progression defined as a greater than 10% decline in the forced vital capacity or death. Measures of safety will include all randomized patients who receive at least one dose of study medication. All adverse events and serious adverse events will be separately tabulated and mapped to a standard classification system and grouped by body system. Any serious adverse events that occur during the trial and 30 days after the end of therapy will be reported to the FDA within 24 hours and followed to outcome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms consistent with IPF with onset between 3 months and 36 months prior to screening
* Worsening as demonstrated by any one of the following within the past year:

  1. >10% decrease in FVC % of predicted,
  2. Worsening chest x-ray or
  3. Worsening dyspnea at rest or on exertion
* Age 20 -79 years of age. Subjects aged 20-50 must have diagnosis by either open or video-assisted thoracic surgery (VATS) lung biopsy
* Diagnosis must be made by (HRCT) showing definite or probable IPF AND either of the following:

  1. Open or VATS lung biopsy showing definite or probable usual interstitial pneumonitis (UIP)
  2. Non-diagnostic transbronchial biopsy to exclude other conditions (including granulomatous disease and malignancies) AND abnormal pulmonary function tests (reduced FVC or decreased DLCO or impaired gas exchange with rest or exercise) AND 2 of the following:

  <!-- -->

  1. Age >50 years
  2. Insidious onset of otherwise unexplained dyspnea or exertion
  3. Bibasilar, inspiratory crackles on examination
* FVC> 55% of predicted value at baseline
* DLCO > 35% of predicted value at screening
* PaO2 >60 mmHg (sea level) or 55 mmHg (altitude) at rest on room air
* Able to understand and willing to provide informed consent prior to any study procedures

Exclusion Criteria:

* History of clinically significant environmental exposure known to cause pulmonary fibrosis
* Diagnosis of connective tissue disease
* FEV1/FVC ratio < 0.6 at screening (post-bronchodilator)
* Residual volume > 120% predicted at screening
* Evidence of active infection
* Any condition other than IPF, which, in the opinion of the site principal investigator, is likely to result in the death of the patient within the next year
* History of unstable or deteriorating cardiac or neurologic disease
* Women with child bearing potential
* Current treatment with corticosteroids, cytoxan, azathioprine, colchicines, pirfenidone, interferon gamma or beta, anti-tumor necrosis factor therapy or with endothelin receptor blockers.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-04; Study Completion 2007-08

PRIMARY OUTCOMES:
Progression defined as a greater than 10% decline in the forced vital capacity (FVC) or death

SECONDARY OUTCOMES:
Change from baseline in % predicted diffusing capacity of the lung for carbon monoxide (DLCO) at 96 weeks
Change from baseline in the resting arterial blood gas (ABG) assessment of A-a gradient at 96 weeks
Change in the number of meters walked in the 6 minute walk test at 96 weeks
Change from baseline in high-resolution computed tomography (HRCT) at 96 weeks
Change from baseline in the quality of life (QOL) assessments
Change in the modified C-reactive protein (CRP) score at 96 weeks
Mortality at 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Craig E Daniels, MD, Principal Investigator — Mayo Clinic; Joseph Lasky, MD, Principal Investigator — Tulane University

REFERENCES:
- [Derived] Daniels CE, Lasky JA, Limper AH, Mieras K, Gabor E, Schroeder DR; Imatinib-IPF Study Investigators. Imatinib treatment for idiopathic pulmonary fibrosis: Randomized placebo-controlled trial results. Am J Respir Crit Care Med. 2010 Mar 15;181(6):604-10. doi: 10.1164/rccm.200906-0964OC. Epub 2009 Dec 10. PMID 20007927
- See also: Related Info — http://www.pulmonaryfibrosis.org/